CLINICAL TRIAL: NCT04777539
Title: Assessing the Safety and Benefit of Home-hospitalization Program in the Management of Natalizumab (Tysabri®) Medication in Multiple Sclerosis
Brief Title: Comparing the Safety and Benefit of Natalizumab (Tysabri®) At-home Infusion vs At-hospital Infusion in Multiple Sclerosis
Acronym: Tys at Home
Status: Active, not recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0442
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis (MS)
Keywords: At-home hospitalization (HAD); Natalizumab; Safety; Medico-economic data; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: At-home natalizumab treated MS patient — MS patient who are treated with natalizumab in at-home hospitalization" (HAD) setting / according at-home hospitalization program

SUMMARY:
At-home use of Natalizumab in multiple sclerosis (MS) patients has been temporarily granted by French security agency of medicines and Health products (ANSM). The main objective of the study is to compare the safety of natalizumab administration at home vs at hospital based on retrospective and prospective data collection. Quality of life, patient perception of at-home natalizumab administration are also evaluated as secondary objectives as well as medico-economic assessment of the method.

Data will be collected for a 12-month retrospective period and a 12-month prospective period.

DETAILED DESCRIPTION:
As part of the Covid-19 pandemic, some neurologists have alerted the French authorities (ANSM: National Medicines Safety Agency) to the interruption of natalizumab treatment by some MS patients. The ANSM has granted temporary home use of natalizumab within the framework of a "at-home hospitalization" (HAD) program. The study purpose is to assess at-home natalizumab administration regarding safety, disease activity, quality of life, patient's perception and costs by comparing outcomes before and after "At Home" natalizumab treatment strategy.

The study consists of two periods of observation: a retrospective one corresponding to the year prior the study entry and a prospective one corresponding to patient follow-up for one year from the date of the patient inclusion. The date of the inclusion corresponds to the natalizumab-infusion conducted at hospital just before infusions hospital at-home started. Retrospective data are collected from medical record and a minimal dataset is needed to enroll the patient regarding MRI activity and safety data (i.e., nature and number of SAE and selected AE of grade 2 the year prior study entry).

The prospective period consists of 10 at-home natalizumab infusions (months 1-5 and 7-11) and 3 at-hospital natalizumab infusions (inclusion, months 6 and 12) according to standard care. In addition to clinical, MRI and safety (SAE and selected AE of grade 2) data collected as part of standard medical care from medical record over all the study period, Quality of life (EQ-5D-5L, MusiQol) and patient's preference (Musicare) questionnaires will be administered at inclusion and months 6 and 12 and clinical global impression of change will be recorded at month 6 and 12. Patients will be asked to notify any adverse events that may occur between each at-home infusion and to record each month his/her healthcare resource consumption in a diary. Patients will be contacted each month after at-home infusion to record safety and healthcare resource consumption data.

For a sub-group of 15 patients qualitative interview will be performed between month 3 and 8 as part of patient preference assessment.

Micro-costing dedicated forms and experts' statements will be used to assess resource utilization associated to natalizumab infusion during each period for medico-analyze purpose.

ELIGIBILITY:
Inclusion Criteria :

1. Male or female over 18 years old;
2. Patients with Relapsing-remitting MS followed in the neurology service
3. Treated for more than 24 months with natalizumab;
4. Anti-JCV negative status at inclusion;
5. Ability to understand the purpose of the study and provide opposition to use protected health information in accordance with national and local subject privacy regulations.
6. Had available medical records to meet study objectives (i.e., SAE and selected AE of grade 2 from the past 12 infusions of natalizumab performed at the hospital before inclusion)
7. Had a cerebral MRI within the previous 12 months (+/- 6 months) which results are available in the medical record.

Exclusion Criteria :

1. Patient having expressed their opposition to the use of their data;
2. Women who are pregnant or breastfeeding or intending to become pregnant during the study;
3. History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic (including diabetes), urologic, pulmonary, neurologic (except for RRMS), dermatologic, psychiatric, renal, or other major disease that would preclude participation in a clinical study, in the opinion of the Investigator.
4. Patient under guardianship or under security measure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with relapsing-remitting MS and treated with natalizumab at hospital will be assessed for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Number of serious Adverse events (SAE) and selected adverse events (AEs) of grade 2 | One year after enrollment
  Grades are based on CTCAE V5. Selected AEs of grade 2: myocarditis, pericarditis, diarrhea, enterocolitis, esophagitis, mucositis, fever/hypothermia folicullitis, papular and/or pustular rash, herpes zoster.

SECONDARY OUTCOMES:
Annualized Relapse Rate | Two time points per patient one year prior to and one year after enrollment
  Annualized Relapse Rate
Change from baseline in T2 lesion load as assessed by MRI | 12-month (+/-6 month) prior enrollment, Baseline (enrollment+/-3 months), 12 months after enrollment
  Modification is based on percentage of patient with at least one new T2 lesion
Change from baseline in gadolinium positive lesion as assessed by MRI | Baseline and 12 month before and 12 month after enrollment
  Modification is based percentage of patient with at least one Gd-enhancing lesion
Multiple Sclerosis International quality of Life (MusiQoL) | Baseline and months 6 and 12
  MusiQoL is a self-administered disease-specific quality of life instrument that comprises 31 items encompassing 9 dimensions: activities of daily living (8), psychological well-being (4), symptoms (3), relationships with friend (4), relationships with family (3), relationship with healthcare system (3), sentimental and sexual life (2), coping (2) and rejection (2). Each item is answered using a 6-point Likert scale (Never/Not at all, Rarely/A little, Sometimes/Somewhat, Often/A lot, Always/Very much and Not applicable)
EuroQol-5Dimension 5Level (EQ-5D-5L) | Baseline and months 6 and 12
  The EQ-5D-5L is a self-administered instrument consisting in 2 components that describe patient's health state:
  A five dimensional questionnaire describing health in terms of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patient is asked to indicate for each one the level of functioning: no problems, slight problems, moderate problems, severe problems and extreme problems.
  A visual analogue scale (VAS) that measures health state (from 0 to 100).
Musicare | Baseline and months 6 and 12
  Musicare is a self-administered disease-specific instrument investigating experience of the quality of care for MS. It comprises 35 items encompassing 5 domains: Information about the disease (11), Information about the treatments/medical investigation (8), Relationships with health care teams (8) Health care access (5) Reception in care structures (3).
Patient experience | One point per patient between months 3 and 8
  Semi-structured interview based on " patient tracer " model will be conducted in a sub-group of 15 patients.
Clinical Global impressions of improvement (CGI-I) | Months 6 and 12
  The CGI is a generic 3-component scale used over the years in a broad range of diseases. The CGI-I (Improvement) is one of the components (one item) measuring change in health state since the entry in the study and can be rated independently.
  CGI-I is rated on a 7-point scale: from 1 (very much improved) to 7 (very much worse).
The average cost per patient | During study, it will be evaluated the average cost per patient for one year of treatment (comparison HDJ vs HAD)
  Compare the cost of the "At home" and "Hospital" management strategies in a before-after design from collective perspective

CONTACTS AND LOCATIONS:
Locations (24):
- France (24):
  - Strasbourg University Hospital, Strasbourg, Bas-Rhin
  - Marseille University Hospital, Marseille, Bouches-du-Rhône
  - Brest University Hospital, Brest, Finistère
  - Quimper Hospital, Quimper, Finistère
  - Bordeaux University Hospital, Bordeaux, Gironde
  - Libourne Hospital, Libourne, Gironde
  - Toulouse University Hospital, Toulouse, Haute-Garonne
  - Limoges University Hospital, Limoges, Haute-Vienne
  - Percy Army Training Hospital, Clamart, Hauts-de-Seine
  - Montpellier University Hospital, Montpellier, Hérault
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Dax Hospital, Dax, Landes
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Orléans Hospital, Orléans, Loiret
  - Lille University Hospital, Lille, Nord
  - Rouen University Hospital, Rouen, Seine-Maritime
  - Poitiers University Hospital, Poitiers, Vienne
  - CH Ajaccio, Ajaccio
  - Les Hôpitaux de Chartres, Chartres
  - CHU Grenoble Alpes, La Tronche
  - Hôpital St Vincent de Paul, Lille
  - Adolphe de Rothschild Ophthalmological Foundation, Paris
  - AP-HP La Pitié-Salpêtrière Hospital, Paris

IPD SHARING:
Plan to Share IPD: No